CLINICAL TRIAL: NCT02372227
Title: A Phase 1 Dose Escalation Study of VS-5584, a Dual PI3K/mTOR Inhibitor, Administered With a Fixed Dose of VS-6063, a Focal Adhesion Kinase Inhibitor, in Subjects With Relapsed Malignant Mesothelioma
Brief Title: A Phase 1 Dose Escalation Study of VS-5584 Administered in Combination With VS-6063, in Subjects With Relapsed Malignant Mesothelioma
Status: Terminated | Phase: Phase 1 | Type: Interventional
Sponsor: Verastem, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: VS-6063-104
Record Dates: First submitted 2015-01-30; First posted 2015-02-26 (Estimated); Last update posted 2017-01-30 (Estimated); Status verified 2017-01

CONDITIONS: Relapsed Malignant Mesothelioma
MeSH Terms: conditions — Mesothelioma, Malignant | interventions — VS-5584; defactinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- VS-5584 and VS-6063 (Experimental)
  Interventions: Drug: VS-5584 and VS-6063

INTERVENTIONS:
Drug: VS-5584 and VS-6063 — Starting dose of VS-5584 will be 20mg taken once daily, 3x/week of each 21 day cycle. All subjects will also receive 2x/day treatment with 400mg VS-6063 in 21 day cycles. Number of Cycles: until progression or unacceptable toxicity develops.

SUMMARY:
The purpose of this study is to evaluate rising dose levels of VS-5584 administered in combination with a fixed dose of VS-6063 in subjects with relapsed malignant mesothelioma to determine a recommended Phase 2 dose (RP2D) for further development of this combination in this indication.

DETAILED DESCRIPTION:
This study is comprised of 2 sequential parts: Part 1 (Dose Escalation of VS-5584) and Part 2 (Expansion). Up to 56 evaluable subjects (i.e., subjects who complete at least 1 cycle [21 days] of therapy) will be enrolled, assuming that:

* Up to 6 dose levels of VS-5584 are studied in Part 1 (Dose Escalation of VS-5584) in combination with a fixed dose of VS-6063 at 400 mg twice daily (BID) with a maximum of 6 subjects enrolled per VS-5584 dose level, for a total of up to 36 subjects (exclusive of replacement subjects).
* Up to an additional 20 evaluable subjects may be enrolled in Part 2, the expansion portion of the study. Subjects will be treated with VS-5584 at the RP2D and schedule determined in the dose escalation portion of the study in combination with a fixed dose of VS-6063.

ELIGIBILITY:
Inclusion Criteria:

1. Histopathologically-confirmed diagnosis of malignant mesothelioma (pleural or peritoneal). Must have disease that has relapsed following at least one prior line of chemotherapy.
2. Must have received at least 3 cycles of first-line chemotherapy.
3. Evaluable or measurable disease as assessed by Response Evaluation Criteria in Solid Tumors (RECIST).
4. Must have archival tumor tissue available for biomarker analysis. A study-specific tumor core biopsy, pleural effusion or ascites sample must be obtained prior to treatment if archival tissue is not available.
5. Performance status according to the Karnofsky Performance Scale ≥70%.
6. Fasting blood glucose of ≤ 140 mg/dL (7.8 mmol/L).
7. Adequate renal function (creatinine ≤ 1.5x upper limit of normal [ULN]) and/or glomerular filtration rate (GFR) of ≥50 mL/min.
8. Adequate hepatic function (total bilirubin ≤ 1.5x ULN; AST and ALT ≤ 3x ULN).
9. Adequate bone marrow function (hemoglobin ≥9.0 g/dL; platelets ≥100 x10^9 cells/L; absolute neutrophil count ≥1.5x10^9 cells/L) without the use of hematopoietic growth factors.

Exclusion Criteria:

1. Have had a previous extra pleural pneumonectomy (EPP).
2. Gastrointestinal condition which could interfere with the swallowing or absorption of study drug.
3. Uncontrolled or severe concurrent medical condition (including uncontrolled brain metastases).
4. Known history of stroke or cerebrovascular accident within 6 months prior to the first dose of study drug.
5. Any evidence of serious active infection.
6. Undergoing active treatment for a secondary malignancy.
7. Cancer-directed therapy (chemotherapy, radiotherapy) within 21 days of the first dose of study drug or 5 half-lives, whichever is shorter.
8. Major surgery within 28 days prior to the first dose of study drug.
9. Acute or chronic pancreatitis.
10. Diabetes mellitus requiring insulin treatment or subjects with a hemoglobin A1C (HbA1C) >7%.
11. History or evidence of cardiac risk.
12. Known history of malignant hypertension.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2015-01; Primary Completion 2015-10 (Actual); Study Completion 2015-10 (Actual)

PRIMARY OUTCOMES:
Incidence of dose-limiting toxicities (DLTs) | 6 months
  Dose Escalation Phase: Frequency of DLTs at each dose level associated with administration of VS-5584 and VS-6063 in a 21 day cycle
Safety and tolerability of the combination of VS-5584 and VS-6063 | 16 months
  Dose Escalation Phase and Expansion Phase: A composite by dose level to include incidence of AEs, SAEs (overall and severity), laboratory abnormalities, ECGs, vital signs, Karnofsky Performance Status, dose interruptions and dose reductions as a measure of safety and tolerability

SECONDARY OUTCOMES:
Pharmacokinetics of VS-5584 & VS-6063 maximum observed plasma concentration (Cmax) | 0-48 hours per patient
Pharmacokinetics of VS-5584 & VS-6063 plasma area under the curve from time zero to last quantifiable concentration (AUClast) | 0-48 hours per patient
Pharmacokinetics of VS-5584 & VS-6063 time to reach maximum observed concentration (Tmax) | 0-48 hours per patient
Pharmacokinetics of VS-5584 & VS-6063 area under the curve from time zero to extrapolated infinite time (AUCO-inf) | 0-48 hours per patient
Pharmacokinetics of VS-5584 & VS-6063 apparent oral clearance (CL/F) | 0-48 hours per patient
Pharmacokinetics of VS-5584 & VS-6063 apparent volume of distribution (Vz/F) | 0-48 hours per patient
Pharmacokinetics of VS-5584 & VS-6063 trough plasma concentration | 0-48 hours per patient

CONTACTS AND LOCATIONS:
Overall Officials: Hagop Youssoufian, Study Chair — Verastem, Inc.
Locations (4):
- United States (2):
  - The University of Chicago Medical Center, Chicago, Illinois
  - Memorial Sloane Kettering Cancer Center, New York, New York
- United Kingdom (2):
  - University of Leicester, Leicester
  - The Institute of Cancer Research, Sutton Surrey